CLINICAL TRIAL: NCT02518646
Title: DElirium prediCtIon in the intenSIve Care Unit: Head to Head comparisON of Two Delirium Prediction Models
Acronym: DECISION
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IC_2015-1782
Record Dates: First submitted 2015-07-21; First posted 2015-08-10 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-01

CONDITIONS: Delirium
Keywords: Delirium; Intensive care unit; Adult; Clinical prediction
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently, two ICU delirium prediction models are available: the PRE-DELIRIC model and the early prediction model (E-PRE-DELRIC). However, the use of these prediction models is not yet implemented as standard in clinical practice, as it is unknown which delirium prediction model can best be used to predict delirium in ICU patients.Therefore the main aim of this study is to compare the performance of the PRE-DELIRIC model and the E-PRE-DELRIC model.

DETAILED DESCRIPTION:
Delirium often occurs in ICU patients and is associated with negative consequences, requiring prevention. A prediction model facilitates the identification of those patients at risk for delirium and therefore need prevention the most. At present, two ICU delirium prediction models are available. First the PRE-DELIRIC model was developed. This recently recalibrated model reliably predicts ICU patients' risk for delirium within 24 hours after ICU admission. Because a relevant number of patients develops delirium during the first 24 hours after ICU admission, and prevention ideally should be deployed as soon as possible, the investigators developed the 'early prediction model' (E-PRE-DELIRIC) which reliably predicts delirium immediately after ICU admission. To implement a delirium prediction model in clinical practice, one needs to know which model best can be used. Currently, the use of a delirium prediction model is not implemented as standard in clinical practice, as this information is unavailable. Therefore the main aim of this study is to compare the (predictive and clinical) performance of the PRE-DELIRIC model and the E-PRE-DELRIC model.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients aged ≥18 years;
* Surgical, medical, neurology/neurosurgical, or trauma patients.

Exclusion Criteria:

* Delirious at ICU admission;
* Expected ICU stay shorter than 6 hours;
* Unable to reliably assess ICU delirium due to:
* sustained coma during entire ICU stay;
* unable to understand the language spoken;
* severely mentally disabled;
* serious receptive aphasia;
* serious auditory or visual disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥ 18 years (surgical, medical, neurology/neurosurgical, or trauma patients) a from the participating multinational ICUs. These ICU patients are at risk of developing the outcome of interest, delirium.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Development of ICU delirium | During the first 14 days after ICU admission
  Defined as a positive assessment for delirium and/or when a patient is treated with haloperidol or other anti-psychotics for delirium (and unable to be assessed).

SECONDARY OUTCOMES:
Delirium subtype | During the first 14 days after ICU admission
  Hyperactive delirium is defined as patients with a persistent positive RASS assessment during the delirium episode (+1 to +4).
  Hypoactive delirium is defined as patients with a persistent neutral or negative RASS assessment during the delirium episode (0 to -3).
  Mixed delirium is defined as patients with both positive and negative RASS assessments during the delirium episode. (Peterson 2006)
Delirium duration | During the first 14 days after ICU admission
  The duration of delirium is defined as time (in days) from the first positive CAM-ICU/ICDSC or treatment with haloperidol or other anti-psychotics for delirium, until the beginning of two consecutive days of negative delirium screenings (negative CAM-ICU/ICDSC).
Delirium episodes | During the first 14 days after ICU admission
  Defined as the number of episodes a patient is screened positive for delirium. A delirium episode is defined as the time from first the positive delirium assessment, until the beginning of two consecutive days (48 hours) of negative delirium assessments.
Delirium onset in a specified period | During the first 14 days after ICU admission
  Based on the quartiles of the time to development of delirium at: day 0-1; day 2; day 3-6; >day 6. These quartiles are based on a former delirium prediction study (E-PRE-DELIRIC). (Wassenaar 2015)
Development of delirium | During the first 14 days after ICU admission
  Defined as ≥ 2 positive assessments for delirium within 48 hours (because of the fluctuating course of delirium).

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, PhD, RN, Principal Investigator — Radboud University Medical Center; Annelies Wassenaar, MSc, RN, Principal Investigator — Radboud University Medical Center; Peter Pickkers, PhD, MD, Principal Investigator — Radboud University Medical Center; Lisette Schoonhoven, PhD, Principal Investigator — University of Southampton
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wassenaar A, van den Boogaard M, van Achterberg T, Slooter AJ, Kuiper MA, Hoogendoorn ME, Simons KS, Maseda E, Pinto N, Jones C, Luetz A, Schandl A, Verbrugghe W, Aitken LM, van Haren FM, Donders AR, Schoonhoven L, Pickkers P. Multinational development and validation of an early prediction model for delirium in ICU patients. Intensive Care Med. 2015 Jun;41(6):1048-56. doi: 10.1007/s00134-015-3777-2. Epub 2015 Apr 18. PMID 25894620
- [Result] van den Boogaard M, Schoonhoven L, Maseda E, Plowright C, Jones C, Luetz A, Sackey PV, Jorens PG, Aitken LM, van Haren FM, Donders R, van der Hoeven JG, Pickkers P. Recalibration of the delirium prediction model for ICU patients (PRE-DELIRIC): a multinational observational study. Intensive Care Med. 2014 Mar;40(3):361-9. doi: 10.1007/s00134-013-3202-7. Epub 2014 Jan 18. PMID 24441670
- [Result] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Derived] van den Boogaard M, Wassenaar A, van Haren FMP, Slooter AJC, Jorens PG, van der Jagt M, Simons KS, Egerod I, Burry LD, Beishuizen A, Pickkers P, Devlin JW. Influence of sedation on delirium recognition in critically ill patients: A multinational cohort study. Aust Crit Care. 2020 Sep;33(5):420-425. doi: 10.1016/j.aucc.2019.12.002. Epub 2020 Feb 5. PMID 32035691
- [Derived] Wassenaar A, Schoonhoven L, Devlin JW, van Haren FMP, Slooter AJC, Jorens PG, van der Jagt M, Simons KS, Egerod I, Burry LD, Beishuizen A, Matos J, Donders ART, Pickkers P, van den Boogaard M. Delirium prediction in the intensive care unit: comparison of two delirium prediction models. Crit Care. 2018 May 5;22(1):114. doi: 10.1186/s13054-018-2037-6. PMID 29728150